CLINICAL TRIAL: NCT07194356
Title: A Randomized Controlled Trial Evaluating the Effect of Preoperative Pericapsular Nerve Group (PENG) Block on Positioning for Spinal Anesthesia and Postoperative Analgesia in Patients Undergoing Hip Fracture Surgery
Brief Title: Effect of Preoperative PENG Block on Spinal Anesthesia Positioning and Postoperative Analgesia in Hip Fracture Surgery
Acronym: PENG-SPINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gülcan GÜL, Specialist in Anesthesiology and Reanimation, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KLKSH-ANES-PENG-001; 2023/514/261/14 (Other: Health Sciences University Kartal Dr. Lutfi Kırdar City Hospital Ethics Committee Approval Number)
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Hip Fractures (ICD-10 72.01-72.2); Postoperative Pain Management After Total Hip Arthroplasty; Elderly Patients; Regional Anesthesia
Keywords: PENG Block; Pericapsular Nerve Group Block; Hip Surgery; Geriatric Anesthesia; Analgesia; Visual Analog Scale; Tramadol; Ultrasound-Guided Block; Positioning Pain; Peripheral Nerve Block
MeSH Terms: conditions — Hip Fractures; Agnosia | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: A randomized, parallel-group, controlled trial evaluating the effectiveness of PENG block versus no block in patients undergoing hip fracture surgery under spinal anesthesia.
Who Masked: Outcomes Assessor
Masking Description: Participants and care providers were not blinded due to the nature of the intervention. However, the outcome assessor who recorded VAS scores and postoperative analgesic consumption was blinded to group assignment to reduce potential bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG Block Group (Experimental): Patients in this group received an ultrasound-guided Pericapsular Nerve Group (PENG) block prior to spinal anesthesia for hip fracture surgery. The block was performed with local anesthetic injection under ultrasound guidance, targeting the articular branches innervating the anterior hip capsule.
  Interventions: Procedure: Pericapsular nerve group (PENG) block
- Control Group (Active Comparator): Patients in this group did not receive a preoperative nerve block. They underwent spinal anesthesia directly for hip fracture surgery without prior intervention. Pain during positioning and postoperative analgesic requirements were evaluated in comparison to the PENG block group.
  Interventions: Procedure: Standard Spinal Anesthesia (Control)

INTERVENTIONS:
Procedure: Pericapsular nerve group (PENG) block — A single-shot PENG block was administered preoperatively using ultrasound guidance. The block was performed with the patient in the supine position, and 20 mL of local anesthetic (0.25% bupivacaine) was injected between the psoas tendon and the superior pubic ramus to achieve analgesia of the anterior hip capsule.
  Arms: PENG Block Group
Procedure: Standard Spinal Anesthesia (Control) — Patients in this arm were managed according to standard care protocols for spinal anesthesia in hip fracture surgery. No preoperative regional block was performed. Pain scores and postoperative tramadol use were measured for comparison with the experimental arm.
  Arms: Control Group

SUMMARY:
Hip fractures are among the most common orthopedic traumas, particularly in elderly patients, and are usually associated with significant pain during positioning for spinal anesthesia. Adequate pain control during positioning can improve patient comfort and facilitate successful administration of anesthesia. The pericapsular nerve group (PENG) block has recently been introduced as a regional anesthesia technique that targets articular branches of the femoral, obturator, and accessory obturator nerves, and has been proposed as a method to reduce pain related to hip fracture positioning.

This study is designed to compare the efficacy of preoperative PENG block versus no block in patients undergoing proximal femoral nailing surgery under spinal anesthesia. The primary objective is to assess its effect on positioning pain using visual analog scale (VAS) scores. Secondary objectives include evaluating its impact on postoperative analgesic consumption, time to first rescue analgesic, and potential side effects.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized controlled trial conducted at the University of Health Sciences, Kartal Dr. Lütfi Kırdar City Hospital. A total of 60 patients, aged 18-90 years, with ASA I-III status, scheduled for proximal femoral nailing (PFN) surgery due to hip fracture, were enrolled. Patients were randomized into two groups using a sealed-envelope method:

PENG Block Group: Received a preoperative ultrasound-guided pericapsular nerve group (PENG) block 30 minutes before spinal anesthesia.

Control Group: Received no block prior to spinal anesthesia.

Standard spinal anesthesia was performed in both groups. All patients received intravenous paracetamol for postoperative analgesia at regular intervals. Additional analgesia with intravenous tramadol was administered if VAS ≥ 4.

The following parameters were collected:

Demographics (age, sex, BMI, ASA status, comorbidities)

Hemodynamic variables (SBP, DBP, HR, SpO₂) at baseline and during perioperative period

VAS scores at baseline, during positioning, and at postoperative time intervals (0, 15, 30 minutes, and 1, 2, 6, 12, and 24 hours)

Time to first rescue analgesic

Total opioid consumption in the first 24 hours postoperatively

Side effects such as nausea, vomiting, or other complications

The study aims to test the hypothesis that PENG block can reduce pain during positioning for spinal anesthesia and may improve postoperative analgesia in patients undergoing hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 90 years

  * ASA (American Society of Anesthesiologists) physical status classification I-III
  * Scheduled for proximal femoral nailing due to hip fracture
  * Able to provide informed consent (or consent provided by a legal representative)
  * Willingness to comply with study procedures and follow-up assessments

Exclusion Criteria:

* - ASA physical status classification IV or V
* Refusal to provide informed consent
* Coagulopathy or current use of anticoagulant therapy contraindicating neuraxial block
* Local infection at the injection site
* Known allergy or hypersensitivity to local anesthetic agents
* Cognitive impairment or inability to cooperate with study procedures
* Severe psychiatric illness preventing reliable pain assessment
* Previous surgery or deformity of the hip interfering with block performance
* Pregnancy or lactation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity during positioning for spinal anesthesia | During spinal anesthesia positioning (within 15 minutes preoperatively)
  Pain scores were recorded using the Visual Analog Scale (VAS; 0-10 cm, where 0 = no pain and 10 = worst pain imaginable) during positioning for spinal anesthesia prior to hip fracture surgery.

SECONDARY OUTCOMES:
Postoperative VAS scores | 0-24 hours after surgery
  Pain scores were assessed using the Visual Analog Scale (VAS) at 2, 6, 12, and 24 hours postoperatively.
Cumulative tramadol requirement in the first 24 hours | 0-24 hours after surgery
  The total dose of intravenous tramadol administered for breakthrough pain was recorded for each patient.
Time to first request for rescue analgesia | 0-24 hours after surgery
  The duration (in hours) between the end of surgery and the first administration of rescue tramadol was recorded.
Incidence of adverse events related to anesthesia | Intraoperative to 24 hours postoperatively
  Frequency of side effects such as nausea, vomiting, hypotension, and local anesthetic systemic toxicity were documented.

CONTACTS AND LOCATIONS:
Overall Officials: Gulcan Gul, M.D., Principal Investigator — Department of Anesthesiology and Reanimation, Kartal Dr. Lütfi Kırdar City Hospital, University of Health Sciences, Istanbul, Turkey
Locations (1):
- Facility Name: Kartal Dr. Lütfi Kırdar City Hospital, University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Plan Description: Individual participant data (IPD) will not be shared because this study was a single-center thesis project with a limited sample size. Only summary-level results and aggregate data will be published in peer-reviewed journals. Patient confidentiality and institutional data protection policies prevent public release of individual-level datasets.